CLINICAL TRIAL: NCT00748761
Title: Cognitive-Behavioral Therapy & Glutamatergic Neurometabolites in Pediatric OCD
Brief Title: Cognitive Behavioral Therapy for Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph O'Neill, PhD, Associate Professor of Child Psychiatry, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH081864 (NIH); R01MH081864 (NIH); DDTR B2-NDO (Other: UCLA)
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; Cognitive-Behavioral Therapy; CBT; MRSI; Glutamate
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Behavior Therapy; Psychotherapy; Waiting Lists; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OCD Active CBT (Experimental): Children with obsessive-compulsive disorder (OCD) will be treated with cognitive behavioral therapy (CBT) from the time of enrollment.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- OCD Waitlist (Active Comparator): Children with OCD will receive waitlist treatment at enrollment. Nonresponders will cross over to CBT.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Waitlist
- Healthy Controls (No Intervention): Healthy control children will be given no intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Nondrug psychotherapy administered weekly for 12 weeks
  Other Names: Behavioral therapy; Psychotherapy; Exposure and response prevention
  Arms: OCD Active CBT; OCD Waitlist
Behavioral: Waitlist — Contact waitlist weekly for 12 weeks
  Other Names: Waiting for treatment; In line for treatment
  Arms: OCD Waitlist

SUMMARY:
This study will examine the way cognitive behavioral therapy changes the structure of the brain in patients with obsessive-compulsive disorder and will thereby determine what makes cognitive behavioral therapy an effective treatment.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) afflicts 2% to 4% of children and adolescents, who suffer from persistent, unwanted thoughts and repetitive behaviors. One of the most effective treatments of OCD is cognitive behavioral therapy (CBT), yet researchers do not know how CBT affects the brain. In this study, brain scans will be performed to determine concentrations of several neurometabolites, which are chemicals involved in providing energy to the brain. Of particular importance are the neurometabolites glutamine and glutamate, which, in addition to providing energy to the brain, are among the most common excitatory neurotransmitters. Disruption of glutamine and glutamate is thought to be related to OCD. By examining where in the brain levels of glutamate and glutamine change, researchers will attempt to determine whether CBT modifies brain activity, whether a circuit targeted by researchers is affected by CBT, and how brain activity in people with OCD differs from that of people without the disorder in terms of the targeted circuit.

Children and adolescents ages 8 through 17 with OCD will be randomly assigned to either receive a 12-week CBT intervention or be placed on a waiting list for 8 weeks before receiving the 12-week intervention. A group of non-OCD participants in the same age group will be used as a control. All groups will undergo magnetic resonance spectroscopic imaging (MRSI), which will measure the concentrations of neurometabolites in multiple brain regions. The control group and the group initially given the CBT intervention will be scanned upon entry of the study and after 12 weeks. The group initially placed on a waiting list will be scanned three times: once upon entry, once after the 8-week waiting period, and once after the 12-week CBT intervention. To determine which participants are benefitting from the treatment, the Yale-Brown Obsessive-Compulsive Scale and other clinical and neurocognitive measures will be administered concurrently with each brain scan.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for OCD as primary diagnosis, based on the Anxiety Disorders Interview Schedule (ADIS) Clinical Severity Rating
* Clinical Global Impressions severity score of at least 4, reflecting moderately ill or worse status
* Children's Yale-Brown Obsessive Compulsive Scale total score of greater than or equal to 16
* No medication for OCD or other psychiatric condition in the past 4 weeks and no use of fluoxetine for the past 6 weeks
* Child is fluent in English
* Parental informed consent and child or adolescent informed assent forms are signed
* For females of childbearing potential a negative pregnancy test will be required for study entry

Exclusion Criteria:

* IQ of less than 80 on the Wechsler Abbreviated Scales of Intelligence
* A lifetime DSM-IV diagnosis of pervasive developmental disorder, mania, psychosis, conduct disorder, or substance dependence assessed through ADIS
* Current DSM-IV diagnosis of major depressive disorder or attention deficit hyperactivity disorder any subtype, assessed through an ADIS rating of 4 or higher
* Any serious psychiatric, psychosocial, or neurological condition, such as a tic disorder, non-OCD anxiety, aggression, or family discord, that requires immediate treatment other than that provided in the current study
* One or more failed adequate trials of exposure-based CBT, defined as at least 10 sessions of therapist-assisted, exposure-based CBT with which the patient voluntarily complied
* More than one failed selective serotonin reuptake inhibitor trial adequate in dose and duration, defined as at least 8 weeks of treatment with at least 20 mg of fluoxetine, 20 mg of paroxetine, 75 mg of sertraline or fluvoxamine, or 75mg of clomipramine
* Any body metal (other than dental fillings), pregnancy, or other contraindications to MRSI scan

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Regional concentration of glutamate and glutamine in brain, as measured by Magnetic Resonance Spectroscopic Imaging (MRSI) | 14 weeks

SECONDARY OUTCOMES:
Overall score on child Yale-Brown Obsessive-Compulsive Scale | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Neill, PhD, Principal Investigator — UCLA Child Psychiatry; John C. Piacentini, PhD, Principal Investigator — UCLA Child Psychiatry
Locations (1):
- UCLA Child Psychiatry, Los Angeles, California, United States